CLINICAL TRIAL: NCT02048384
Title: An Exploratory Study of Metformin With or Without Rapamycin as Maintenance Therapy After Induction Chemotherapy in Subjects With Metastatic Pancreatic Adenocarcinoma
Brief Title: A Study of Metformin With or Without Rapamycin as Maintenance Therapy After Induction Chemotherapy in Subjects With Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Stand Up To Cancer (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J13146; NA_00090282 (Other: JHMIRB)
Record Dates: First submitted 2014-01-23; First posted 2014-01-29 (Estimated); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
Keywords: rapamycin; metformin; pancreatic cancer; adenocarcinoma; metastatic
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma; Neoplasm Metastasis | interventions — Metformin; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A - metformin alone (Experimental): metformin alone Arm A patients will receive metformin 850mg orally twice a day on a 28 day cycle.
  Interventions: Drug: metformin alone (Arm A)
- B - metformin + rapamycin (Active Comparator): metformin + rapamycin Arm B patients will receive 850mg orally twice a day and rapamycin 4mg orally once a day on a 28 day cycle.
  Interventions: Drug: metformin (Arm B); Drug: rapamycin (Arm B)

INTERVENTIONS:
Drug: metformin alone (Arm A) — metformin alone
  Other Names: Glumetza, Fortamet, Riomet, Glucophage
  Arms: A - metformin alone
Drug: metformin (Arm B) — rapamycin + metformin
  Other Names: Glumetza, Fortamet, Riomet, Glucophage
  Arms: B - metformin + rapamycin
Drug: rapamycin (Arm B) — rapamycin + metformin
  Other Names: Sirolimus, Rapamune
  Arms: B - metformin + rapamycin

SUMMARY:
This is a phase 1b, multi-center, open label, randomized study to evaluate the safety and feasibility of administering metformin with or without rapamycin after disease stabilization on chemotherapy in subjects with metastatic PDA.

DETAILED DESCRIPTION:
Subjects with metastatic PDA who have received FOLFIRINOX or a gemcitabine-containing regimen and have achieved stable disease or better will be enrolled onto this study. Subjects should have had at least 6 months of chemotherapy and decline continuation of chemotherapy and should have stable disease or better on 2 scans taken at least 6 weeks apart. If applicable, subjects should also have a stable or declining CA19-9.

Twenty-two subjects will be randomized in a 1:1 ratio to metformin (Arm A) or metformin + rapamycin (Arm B). Subjects will be stratified according to their prior chemotherapy regimen: FOLFIRINOX or a gemcitabine-containing regimen.

Treatments will be administered orally on a 28 day cycle. Metformin will be administered 850mg twice daily and rapamycin will be administered 4mg daily.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic pancreatic adenocarcinoma. Subjects with islet cell neoplasms are excluded.
* Have received 6 months of chemotherapy.
* Have stable disease for at least 6 months on the current regimen with the last 2 scans taken at least 6 months apart. Measurable disease not required.
* Eastern Cooperative Oncology Group performance status 0 or 1.
* Life expectancy of greater than 12 weeks.
* Adequate organ and marrow function.
* Oxygen saturation on room air > 92 % by pulse oximetry. (Subjects on intermittent or continuous supplemental oxygen are excluded).
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Receiving or has received any other investigational agents within 28 days prior to Day 1 of treatment in this study.
* Has undergone major surgery, other than diagnostic surgery (i.e. surgery done to obtain a biopsy for diagnosis or an aborted Whipple), within 28 days prior to Day 1 of treatment in this study.
* Known history of brain metastases unless previously treated and well controlled for at least 3 months (defined as stable clinically, no edema, no steroids).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to metformin or rapamycin.
* Taking ketoconazole, voriconazole, itraconazole, erythromycin, telithromycin, clarithromycin, rifampin, rifabutin, bromocriptine, cimetidine, cisapride, clotrimazole, danazol, diltiazem, fluconazole, protease inhibitors (e.g., HIV and hepatitis C that include drugs such as ritonavir, indinavir, boceprevir, and telaprevir), metoclopramide, nicardipine, troleandomycin, verapamil, carbamazepine, phenobarbital, phenytoin, rifapentine, St. John's Wort (Hypericum perforatum), and grapefruit juice. Subjects on metformin will not be excluded.
* Has received any non-oncology live vaccine therapy used for prevention of infectious diseases for up to 28 days prior to or after the initiation of treatment in this study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (bacterial, viral, or fungal infection(s) requiring systemic therapy), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Has serious medical risk factors involving any of the major organ systems such that the Investigator considers it unsafe for the subject to receive an experimental research drug.
* Unhealed surgical wound or other clinically significant wound.
* Known history of chronic HIV, Hepatitis B or hepatitis C infections.
* Pregnant or breast feeding.
* Unwilling or unable to comply with study procedures.
* Cannot reliably swallow pills.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-06-10 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
safety and feasibility | 1 year
  To determine the safety and feasibility of administering metformin with or without rapamycin in subjects with metastatic pancreatic ductal adenocarcinoma (PDA) after disease stabilization on chemotherapy.

OTHER OUTCOMES:
FDG uptake | 1 year
  To evaluate fludeoxyglucose (FDG) uptake in metastatic PDA subjects treated with metformin with or without rapamycin.
mTOR activity | 1 year
  To measure mammalian target of rapamycin (mTOR) activity in peripheral blood mononuclear cells (PBMC) of subjects treated with metformin with or without rapamycin.
estimation of RR, TTP, PFS, OS | 1 year
  To estimate response rate (RR), time to progression (TTP), progression-free survival (PFS) and overall survival (OS) in subjects with metastatic PDA treated with metformin with or without rapamycin.
CA19-9 measurement | 1 year
  To measure tumor marker kinetics (CA 19-9) in subjects treated with metformin with or without rapamycin.

CONTACTS AND LOCATIONS:
Overall Officials: Dung Le, MD, Study Chair — Johns Hopkins SKCCC
Locations (2):
- United States (2):
  - Scottsdale Healthcare Hospitals DBA Honor Health, Scottsdale, Arizona
  - Johns Hopkins SKCCC, Baltimore, Maryland